CLINICAL TRIAL: NCT01706939
Title: The Quarterback Trial: A Randomized Phase III Clinical Trial Comparing Reduced and Standard Radiation Therapy Doses for Locally Advanced HPV Positive Oropharynx Cancer
Brief Title: The Quarterback Trial: Reduced Dose Radiotherapy for HPV+ Oropharynx Cancer
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Collaborators: Biodesign Institute (Other); Arizona State University (Other)
Responsible Party: Principal Investigator, Marshall Posner, MD, Director, Head and Neck Medical Oncology, Icahn School of Medicine at Mount Sinai
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GCO 12-1050
Record Dates: First submitted 2012-09-14; First posted 2012-10-15 (Estimated); Results first posted 2022-09-01 (Actual); Last update posted 2024-08-29 (Actual); Status verified 2024-08

CONDITIONS: Squamous Cell Carcinomas
Keywords: Reduced radiotherapy; Randomization, Phase III; Reduced radiation therapy; head and neck; oropharynx; unknown primary (cervical lymph nodes); nasopharynx primary; HPV; p16
MeSH Terms: conditions — Carcinoma, Squamous Cell | interventions — Radiation; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Reduced Dose Radiation (Experimental): Patients randomized to receive a reduced (5600 cGy) dose radiotherapy with weekly Carboplatin
  Interventions: Radiation: Reduced Dose Radiation; Drug: Carboplatin
- Standard Dose Radiation (Active Comparator): Patients randomized to receive a standard (7000 cGy) dose radiotherapy with carboplatin
  Interventions: Radiation: Standard Dose Radiation; Drug: Carboplatin

INTERVENTIONS:
Radiation: Reduced Dose Radiation — Reduced Dose Radiation (5600 cGy) dose radiotherapy
  Arms: Reduced Dose Radiation
Radiation: Standard Dose Radiation — Standard Dose Radiation (7000 cGy) dose radiotherapy
  Arms: Standard Dose Radiation
Drug: Carboplatin — Day 1, every 7 days ( + 2 days)

SUMMARY:
This trial aims to directly compare a reduced radiation dose to the standard of care in HPVOPC for non-inferiority, thus allowing for direct comparison of outcomes between the two groups. The study hypothesis is that LRC and PFS at 3 years for reduced dose CRT are non-inferior to standard dose CRT.

DETAILED DESCRIPTION:
This is a randomized Phase III study comparing two doses of definitive radiation therapy given with induction and concurrent chemotherapy in HPV-positive oropharynx, unknown primary or nasopharynx cancer. Eligible, consented and registered patients will receive three cycles of Docetaxel Cisplatin and 5-FU (TPF) induction chemotherapy. After 3 cycles, the patients will be assessed for clinical, radiographic and pathologic response to TPF. Patients with a clinical or radiographic CR or PR will be randomized on the second phase of this study, where patients will undergo a 2:1 randomization to reduced (5600 cGy) or standard (7000 cGy) dose radiotherapy with weekly Carboplatin. Patients not meeting the response criteria will be treated with standard dose CRT. Patients not completing 3 cycles TPF for reasons of toxicity, progressive disease, choice, or other medical necessity will be treated with standard dose CRT or surgery depending on their primary site and overall medical condition and followed for survival. Toxicity will be assessed by Symptom scores, QOL and SAE monitoring. The primary end point of the trial is equivalent local regional control and PFS at 3 years. Patients will be followed for 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have histologically or cytologically confirmed squamous cell carcinoma of the oropharynx, unknown primary, or nasopharynx that is HPV positive as determined by PCR and p16 positive as determined by IHC. Tissue from the primary site must be available for biomarker studies. PCR and IHC must be performed in the central laboratory (Zhang, MSSM)
* Stage 3 or 4 disease without evidence of distant metastases.
* At least one clinically evaluable or uni- or bi-dimensionally measurable lesion by RECIST 1.1 criteria.
* Age > 18 years.
* No previous surgery, radiation therapy or chemotherapy for SSCHN (other than biopsy or tonsillectomy) is allowed at time of study entry.
* ECOG performance status of 0 or 1.
* No active alcohol addiction (as assessed by medical caregiver and defined as at least 6 months without activity).
* Participants must have adequate bone marrow, hepatic and renal functions as defined in the protocol.
* Ability to understand and the willingness to sign a written informed consent document.
* Patients with Gilbert's Disease and absent hepatic pathology by history and clinical assessment maybe treated on study with bilirubins > the ULN for the institution if other liver function studies are within the normal range

Exclusion Criteria:

* Pregnant or breast feeding women, or women and men of childbearing potential not willing to use adequate contraception while on treatment and for at least 3 months thereafter.
* Previous or current malignancies at other sites, with the exception of adequately treated in situ carcinoma of the cervix, basal or squamous cell carcinoma of the skin, thyroid cancer, or other cancer curatively treated by surgery and with no current evidence of disease for at least 5 years.
* Symptomatic peripheral neuropathy ≥ grade 2 by NCI Common Terminology Criteria (NCI-CTC) version 4.
* Symptomatic altered hearing > grade 2 by NCI-CTCv4 criteria.
* Other serious illnesses or medical conditions including but not limited to:

  1. Unstable cardiac disease despite treatment, myocardial infarction within 6 months prior to study entry
  2. History of significant neurologic or psychiatric disorders including dementia or seizures
  3. Active clinically significant uncontrolled infection
  4. Active peptic ulcer disease defined as unhealed or clinically active
  5. Hypercalcemia
  6. Active drug addiction including alcohol, cocaine or intravenous drug use defined as occurring within the 6 months preceding diagnosis
  7. Chronic Obstructive Pulmonary Disease, defined as being associated with a hospitalization for pneumonia or respiratory decompensation within 12 months of diagnosis. This does not include obstruction from tumor
  8. Autoimmune disease requiring therapy, prior organ transplant, or HIV infection
  9. Interstitial lung disease
  10. Hepatitis C (test required)
* Patients that have experienced an involuntary weight loss of more than 25% of their body weight in the 2 months preceding study entry.
* Concurrent treatment with any other anticancer therapy.
* Participation in an investigational therapeutic drug trial within 30 days of study entry.
* Active smoking within the past 20 years with a cumulative Pack Year history of > 20 Pack Years or active smoking (Defined as > 1 cigarette per day) within the last 2 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2012-09-01 (Actual); Primary Completion 2020-04-01 (Actual); Study Completion 2035-05-01 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Marshall Posner, M.D., Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided
randomized trial should not be shared until trial is over.

REFERENCES:
- [Background] Chaturvedi AK, Engels EA, Pfeiffer RM, Hernandez BY, Xiao W, Kim E, Jiang B, Goodman MT, Sibug-Saber M, Cozen W, Liu L, Lynch CF, Wentzensen N, Jordan RC, Altekruse S, Anderson WF, Rosenberg PS, Gillison ML. Human papillomavirus and rising oropharyngeal cancer incidence in the United States. J Clin Oncol. 2011 Nov 10;29(32):4294-301. doi: 10.1200/JCO.2011.36.4596. Epub 2011 Oct 3. PMID 21969503
- [Background] Chaturvedi AK, Engels EA, Anderson WF, Gillison ML. Incidence trends for human papillomavirus-related and -unrelated oral squamous cell carcinomas in the United States. J Clin Oncol. 2008 Feb 1;26(4):612-9. doi: 10.1200/JCO.2007.14.1713. PMID 18235120
- [Background] Nasman A, Attner P, Hammarstedt L, Du J, Eriksson M, Giraud G, Ahrlund-Richter S, Marklund L, Romanitan M, Lindquist D, Ramqvist T, Lindholm J, Sparen P, Ye W, Dahlstrand H, Munck-Wikland E, Dalianis T. Incidence of human papillomavirus (HPV) positive tonsillar carcinoma in Stockholm, Sweden: an epidemic of viral-induced carcinoma? Int J Cancer. 2009 Jul 15;125(2):362-6. doi: 10.1002/ijc.24339. PMID 19330833
- [Background] Andl T, Kahn T, Pfuhl A, Nicola T, Erber R, Conradt C, Klein W, Helbig M, Dietz A, Weidauer H, Bosch FX. Etiological involvement of oncogenic human papillomavirus in tonsillar squamous cell carcinomas lacking retinoblastoma cell cycle control. Cancer Res. 1998 Jan 1;58(1):5-13. PMID 9426048
- [Background] Munger K, Baldwin A, Edwards KM, Hayakawa H, Nguyen CL, Owens M, Grace M, Huh K. Mechanisms of human papillomavirus-induced oncogenesis. J Virol. 2004 Nov;78(21):11451-60. doi: 10.1128/JVI.78.21.11451-11460.2004. No abstract available. PMID 15479788
- [Background] Psyrri A, DeFilippis RA, Edwards AP, Yates KE, Manuelidis L, DiMaio D. Role of the retinoblastoma pathway in senescence triggered by repression of the human papillomavirus E7 protein in cervical carcinoma cells. Cancer Res. 2004 May 1;64(9):3079-86. doi: 10.1158/0008-5472.can-03-3739. PMID 15126344
- [Background] Weinberger PM, Yu Z, Haffty BG, Kowalski D, Harigopal M, Brandsma J, Sasaki C, Joe J, Camp RL, Rimm DL, Psyrri A. Molecular classification identifies a subset of human papillomavirus--associated oropharyngeal cancers with favorable prognosis. J Clin Oncol. 2006 Feb 10;24(5):736-47. doi: 10.1200/JCO.2004.00.3335. Epub 2006 Jan 9. PMID 16401683
- [Background] Ang KK, Harris J, Wheeler R, Weber R, Rosenthal DI, Nguyen-Tan PF, Westra WH, Chung CH, Jordan RC, Lu C, Kim H, Axelrod R, Silverman CC, Redmond KP, Gillison ML. Human papillomavirus and survival of patients with oropharyngeal cancer. N Engl J Med. 2010 Jul 1;363(1):24-35. doi: 10.1056/NEJMoa0912217. Epub 2010 Jun 7. PMID 20530316
- [Background] Gillison ML, Koch WM, Capone RB, Spafford M, Westra WH, Wu L, Zahurak ML, Daniel RW, Viglione M, Symer DE, Shah KV, Sidransky D. Evidence for a causal association between human papillomavirus and a subset of head and neck cancers. J Natl Cancer Inst. 2000 May 3;92(9):709-20. doi: 10.1093/jnci/92.9.709. PMID 10793107
- [Background] Gillison ML. Human papillomavirus and prognosis of oropharyngeal squamous cell carcinoma: implications for clinical research in head and neck cancers. J Clin Oncol. 2006 Dec 20;24(36):5623-5. doi: 10.1200/JCO.2006.07.1829. No abstract available. PMID 17179099
- [Background] Ringstrom E, Peters E, Hasegawa M, Posner M, Liu M, Kelsey KT. Human papillomavirus type 16 and squamous cell carcinoma of the head and neck. Clin Cancer Res. 2002 Oct;8(10):3187-92. PMID 12374687
- [Background] Lassen P, Eriksen JG, Hamilton-Dutoit S, Tramm T, Alsner J, Overgaard J. Effect of HPV-associated p16INK4A expression on response to radiotherapy and survival in squamous cell carcinoma of the head and neck. J Clin Oncol. 2009 Apr 20;27(12):1992-8. doi: 10.1200/JCO.2008.20.2853. Epub 2009 Mar 16. PMID 19289615
- [Background] Licitra L, Perrone F, Bossi P, Suardi S, Mariani L, Artusi R, Oggionni M, Rossini C, Cantu G, Squadrelli M, Quattrone P, Locati LD, Bergamini C, Olmi P, Pierotti MA, Pilotti S. High-risk human papillomavirus affects prognosis in patients with surgically treated oropharyngeal squamous cell carcinoma. J Clin Oncol. 2006 Dec 20;24(36):5630-6. doi: 10.1200/JCO.2005.04.6136. PMID 17179101
- [Background] Cmelak AJ, Li S, Goldwasser MA, Murphy B, Cannon M, Pinto H, Rosenthal DI, Gillison M, Forastiere AA. Phase II trial of chemoradiation for organ preservation in resectable stage III or IV squamous cell carcinomas of the larynx or oropharynx: results of Eastern Cooperative Oncology Group Study E2399. J Clin Oncol. 2007 Sep 1;25(25):3971-7. doi: 10.1200/JCO.2007.10.8951. PMID 17761982
- [Background] Fakhry C, Westra WH, Li S, Cmelak A, Ridge JA, Pinto H, Forastiere A, Gillison ML. Improved survival of patients with human papillomavirus-positive head and neck squamous cell carcinoma in a prospective clinical trial. J Natl Cancer Inst. 2008 Feb 20;100(4):261-9. doi: 10.1093/jnci/djn011. Epub 2008 Feb 12. PMID 18270337
- [Background] Worden FP, Kumar B, Lee JS, Wolf GT, Cordell KG, Taylor JM, Urba SG, Eisbruch A, Teknos TN, Chepeha DB, Prince ME, Tsien CI, D'Silva NJ, Yang K, Kurnit DM, Mason HL, Miller TH, Wallace NE, Bradford CR, Carey TE. Chemoselection as a strategy for organ preservation in advanced oropharynx cancer: response and survival positively associated with HPV16 copy number. J Clin Oncol. 2008 Jul 1;26(19):3138-46. doi: 10.1200/JCO.2007.12.7597. Epub 2008 May 12. PMID 18474879
- [Background] Rischin D, Young RJ, Fisher R, Fox SB, Le QT, Peters LJ, Solomon B, Choi J, O'Sullivan B, Kenny LM, McArthur GA. Prognostic significance of p16INK4A and human papillomavirus in patients with oropharyngeal cancer treated on TROG 02.02 phase III trial. J Clin Oncol. 2010 Sep 20;28(27):4142-8. doi: 10.1200/JCO.2010.29.2904. Epub 2010 Aug 9. PMID 20697079
- [Background] Lorch JH, Goloubeva O, Haddad RI, Cullen K, Sarlis N, Tishler R, Tan M, Fasciano J, Sammartino DE, Posner MR; TAX 324 Study Group. Induction chemotherapy with cisplatin and fluorouracil alone or in combination with docetaxel in locally advanced squamous-cell cancer of the head and neck: long-term results of the TAX 324 randomised phase 3 trial. Lancet Oncol. 2011 Feb;12(2):153-9. doi: 10.1016/S1470-2045(10)70279-5. Epub 2011 Jan 11. PMID 21233014
- [Background] Posner MR, Lorch JH, Goloubeva O, Tan M, Schumaker LM, Sarlis NJ, Haddad RI, Cullen KJ. Survival and human papillomavirus in oropharynx cancer in TAX 324: a subset analysis from an international phase III trial. Ann Oncol. 2011 May;22(5):1071-1077. doi: 10.1093/annonc/mdr006. Epub 2011 Feb 11. PMID 21317223
- [Background] Machtay M, Moughan J, Trotti A, Garden AS, Weber RS, Cooper JS, Forastiere A, Ang KK. Factors associated with severe late toxicity after concurrent chemoradiation for locally advanced head and neck cancer: an RTOG analysis. J Clin Oncol. 2008 Jul 20;26(21):3582-9. doi: 10.1200/JCO.2007.14.8841. Epub 2008 Jun 16. PMID 18559875
- [Background] Adelstein DJ, Li Y, Adams GL, Wagner H Jr, Kish JA, Ensley JF, Schuller DE, Forastiere AA. An intergroup phase III comparison of standard radiation therapy and two schedules of concurrent chemoradiotherapy in patients with unresectable squamous cell head and neck cancer. J Clin Oncol. 2003 Jan 1;21(1):92-8. doi: 10.1200/JCO.2003.01.008. PMID 12506176
- [Background] Forastiere A, Maor M, Weber R, Pajak, T, Glisson B, Trotti A, Ridge J, et al. Long term results of Intergroup RTOG 91-11: A Phase III trial to preserve the larynx - Induction cisplatin/5-FU and radiation therapy versus concurrent cisplatin and radiation therapy versus radiation therapy. Proceedings of the American Society of Clinical Oncology. 2006:5517.
- [Background] Staar S, Rudat V, Stuetzer H, Dietz A, Volling P, Schroeder M, Flentje M, Eckel HE, Mueller RP. Intensified hyperfractionated accelerated radiotherapy limits the additional benefit of simultaneous chemotherapy--results of a multicentric randomized German trial in advanced head-and-neck cancer. Int J Radiat Oncol Biol Phys. 2001 Aug 1;50(5):1161-71. doi: 10.1016/s0360-3016(01)01544-9. PMID 11483325
- [Background] Taylor SG 4th, Murthy AK, Vannetzel JM, Colin P, Dray M, Caldarelli DD, Shott S, Vokes E, Showel JL, Hutchinson JC, et al. Randomized comparison of neoadjuvant cisplatin and fluorouracil infusion followed by radiation versus concomitant treatment in advanced head and neck cancer. J Clin Oncol. 1994 Feb;12(2):385-95. doi: 10.1200/JCO.1994.12.2.385. PMID 8113846
- [Background] Best SR, Ha PK, Blanco RG, Saunders JR Jr, Zinreich ES, Levine MA, Pai SI, Walker M, Trachta J, Ulmer K, Murakami P, Thompson R, Califano JA, Messing BP. Factors associated with pharyngoesophageal stricture in patients treated with concurrent chemotherapy and radiation therapy for oropharyngeal squamous cell carcinoma. Head Neck. 2011 Dec;33(12):1727-34. doi: 10.1002/hed.21657. Epub 2011 Jan 18. PMID 21246640
- [Background] Bonner JA, Harari PM, Giralt J, Cohen RB, Jones CU, Sur RK, Raben D, Baselga J, Spencer SA, Zhu J, Youssoufian H, Rowinsky EK, Ang KK. Radiotherapy plus cetuximab for locoregionally advanced head and neck cancer: 5-year survival data from a phase 3 randomised trial, and relation between cetuximab-induced rash and survival. Lancet Oncol. 2010 Jan;11(1):21-8. doi: 10.1016/S1470-2045(09)70311-0. Epub 2009 Nov 10. PMID 19897418
- [Background] Agoston ES, Robinson SJ, Mehra KK, Birch C, Semmel D, Mirkovic J, Haddad RI, Posner MR, Kindelberger D, Krane JF, Brodsky J, Crum CP. Polymerase chain reaction detection of HPV in squamous carcinoma of the oropharynx. Am J Clin Pathol. 2010 Jul;134(1):36-41. doi: 10.1309/AJCP1AAWXE5JJCLZ. PMID 20551264
- [Background] Harris SL, Thorne LB, Seaman WT, Hayes DN, Couch ME, Kimple RJ. Association of p16(INK4a) overexpression with improved outcomes in young patients with squamous cell cancers of the oral tongue. Head Neck. 2011 Nov;33(11):1622-7. doi: 10.1002/hed.21650. Epub 2010 Dec 28. PMID 21990227
- [Background] Schache AG, Liloglou T, Risk JM, Filia A, Jones TM, Sheard J, Woolgar JA, Helliwell TR, Triantafyllou A, Robinson M, Sloan P, Harvey-Woodworth C, Sisson D, Shaw RJ. Evaluation of human papilloma virus diagnostic testing in oropharyngeal squamous cell carcinoma: sensitivity, specificity, and prognostic discrimination. Clin Cancer Res. 2011 Oct 1;17(19):6262-71. doi: 10.1158/1078-0432.CCR-11-0388. PMID 21969383
- [Background] Maxwell JH, Kumar B, Feng FY, Worden FP, Lee JS, Eisbruch A, Wolf GT, Prince ME, Moyer JS, Teknos TN, Chepeha DB, McHugh JB, Urba SG, Stoerker J, Walline HM, Kurnit DM, Cordell KG, Davis SJ, Ward PD, Bradford CR, Carey TE. Tobacco use in human papillomavirus-positive advanced oropharynx cancer patients related to increased risk of distant metastases and tumor recurrence. Clin Cancer Res. 2010 Feb 15;16(4):1226-35. doi: 10.1158/1078-0432.CCR-09-2350. Epub 2010 Feb 9. PMID 20145161
- [Background] Anderson KS, Wong J, D'Souza G, Riemer AB, Lorch J, Haddad R, Pai SI, Longtine J, McClean M, LaBaer J, Kelsey KT, Posner M. Serum antibodies to the HPV16 proteome as biomarkers for head and neck cancer. Br J Cancer. 2011 Jun 7;104(12):1896-905. doi: 10.1038/bjc.2011.171. PMID 21654689
- [Background] Kumar B, Cordell KG, Lee JS, Worden FP, Prince ME, Tran HH, Wolf GT, Urba SG, Chepeha DB, Teknos TN, Eisbruch A, Tsien CI, Taylor JM, D'Silva NJ, Yang K, Kurnit DM, Bauer JA, Bradford CR, Carey TE. EGFR, p16, HPV Titer, Bcl-xL and p53, sex, and smoking as indicators of response to therapy and survival in oropharyngeal cancer. J Clin Oncol. 2008 Jul 1;26(19):3128-37. doi: 10.1200/JCO.2007.12.7662. Epub 2008 May 12. PMID 18474878
- [Background] Porceddu SV, Pryor DI, Burmeister E, Burmeister BH, Poulsen MG, Foote MC, Panizza B, Coman S, McFarlane D, Coman W. Results of a prospective study of positron emission tomography-directed management of residual nodal abnormalities in node-positive head and neck cancer after definitive radiotherapy with or without systemic therapy. Head Neck. 2011 Dec;33(12):1675-82. doi: 10.1002/hed.21655. Epub 2011 Jan 14. PMID 22076976
- [Background] Riemer AB, Keskin DB, Zhang G, Handley M, Anderson KS, Brusic V, Reinhold B, Reinherz EL. A conserved E7-derived cytotoxic T lymphocyte epitope expressed on human papillomavirus 16-transformed HLA-A2+ epithelial cancers. J Biol Chem. 2010 Sep 17;285(38):29608-22. doi: 10.1074/jbc.M110.126722. Epub 2010 Jul 8. PMID 20615877
- [Derived] Takahashi M, Hwang M, Misiukiewicz K, Gupta V, Miles BA, Bakst R, Genden E, Selkridge I, Botzler J, Virani V, Moshier E, Bonomi MR, Posner MR. Quality of Life Analysis of HPV-Positive Oropharyngeal Cancer Patients in a Randomized Trial of Reduced-Dose Versus Standard Chemoradiotherapy: 5-Year Follow-Up. Front Oncol. 2022 Apr 8;12:859992. doi: 10.3389/fonc.2022.859992. eCollection 2022. PMID 35463348
- [Derived] Psyrri A, Rampias T, Vermorken JB. The current and future impact of human papillomavirus on treatment of squamous cell carcinoma of the head and neck. Ann Oncol. 2014 Nov;25(11):2101-2115. doi: 10.1093/annonc/mdu265. Epub 2014 Jul 23. PMID 25057165

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 23 participants were assessed and started in pre-randomization induction phase. Participants were not randomized until after they completed the pre-randomization phase and TPF induction.
Groups:
- Pre-Randomization: Participants received three cycles of Docetaxel, Cisplatin and 5-RU (TPF)
- Reduced Dose Radiation: After TPF induction chemotherapy patients randomized to receive a reduced (5600 cGy) dose radiotherapy with weekly Carboplatin
  Reduced Dose Radiation: Reduced Dose Radiation (5600 cGy) dose radiotherapy
  Carboplatin: Day 1, every 7 days ( + 2 days)
- Standard Dose Radiation: After TPF induction chemotherapy patients randomized to receive a standard (7000 cGy) dose radiotherapy with carboplatin
  Standard Dose Radiation: Standard Dose Radiation (7000 cGy) dose radiotherapy
  Carboplatin: Day 1, every 7 days ( + 2 days)
Period: Pre Randomization
Arm/Group | Pre-Randomization | Reduced Dose Radiation | Standard Dose Radiation
Started | 23 | 0 | 0
Completed | 20 | 0 | 0
Not Completed | 3 | 0 | 0
Not completed — Screen Failure | 1 | 0 | 0
Not completed — Ineligible for Randomization | 1 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0
Period: Randomization
Arm/Group | Pre-Randomization | Reduced Dose Radiation | Standard Dose Radiation
Started | 0 | 12 | 8
Completed | 0 | 9 | 6
Not Completed | 0 | 3 | 2
Not completed — Insufficient QoL survey compliance | 0 | 1 | 1
Not completed — Progression of disease | 0 | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Reduced Dose Radiation | Standard Dose Radiation | Total
Number analyzed (Participants) | 12 | 8 | 20
Age, Continuous [Median (Full Range); unit: years] | 55 [36 to 78] | 57 [36 to 78] | 56.5 [36 to 78]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 1
  Male | 11 | 8 | 19
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 2
  Not Hispanic or Latino | 11 | 7 | 18
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 2 | 6
  White | 8 | 6 | 14
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Tumor Site [Count of Participants; unit: Participants]
  Base of Tongue (BOT) | 5 | 5 | 10
  Tonsil | 7 | 3 | 10
HPV Status [Count of Participants; unit: Participants]
  HPV 16 | 10 | 6 | 16
  Other than HPV 16 | 2 | 2 | 4
Smoking Status [Count of Participants; unit: Participants]
  Never smoker | 9 | 3 | 12
  <10 pack-years | 3 | 2 | 5
  10-20 pack-years | 0 | 3 | 3

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Progression Free Survival (PFS)
Description: Progression free survival (PFS) at 5 years in patients with advanced HPV related oropharynx cancer, nasopharynx cancer or unknown primary treated with reduced or standard dose radiation.
Time Frame: at 3 and 5 years
Measure: Count of Participants; unit: Participants
Arm/Group | Reduced Dose Radiation | Standard Dose Radiation
Number analyzed (Participants) | 12 | 8
Participants
  at 3 years | 10 | 7
  at 5 years | 10 | 7

2. Secondary Outcome: Number of Participants With Local-regional Control
Description: Local-regional control (LRC) at 3 years in patients with advanced HPV related oropharynx cancer or unknown primary treated with reduced or standard dose radiation.
Time Frame: at 3 years
Measure: Count of Participants; unit: Participants
Arm/Group | Reduced Dose Radiation | Standard Dose Radiation
Number analyzed (Participants) | 12 | 8
Participants | 10 | 7

3. Secondary Outcome: Number of Participants With Overall Survival at 5 Years
Description: Overall Survival (OS) 5 years treated with reduced or standard dose CRT.
Time Frame: at 5 years
Measure: Count of Participants; unit: Participants
Arm/Group | Reduced Dose Radiation | Standard Dose Radiation
Number analyzed (Participants) | 12 | 8
Participants | 10 | 7

4. Secondary Outcome: Number of Participants With Acute Toxicity of Chemoradiotherapy (CRT)
Description: Number of participants with acute toxicity treated with reduced or standard dose CRT.
Time Frame: at 5 years
Measure: Count of Participants; unit: Participants
Arm/Group | Reduced Dose Radiation | Standard Dose Radiation
Number analyzed (Participants) | 12 | 8
Participants | 3 | 1

5. Secondary Outcome: Biomarkers Predictive of Failure
Description: To determine biomarkers predictive of failure with either reduced or standard dose radiotherapy.
Time Frame: at 5 years
Measure: Number; unit: biomarkers
Arm/Group | Reduced Dose Radiation | Standard Dose Radiation
Number analyzed (Participants) | 12 | 8
biomarkers | 0 | 0

6. Secondary Outcome: Overall Survival at 15 Years
Time Frame: at 15 years
Reporting Status: Not Posted, anticipated posting 2035-05

7. Secondary Outcome: Change in MD Anderson Dysphagia Inventory (MDADI) From Baseline
Description: MDADI is a questionnaire of 20 questions and contains a global subscale, and three other categories of questions (emotional, functional, and physical). The scores are summed and a mean score is calculated. This mean score was multiplied by 20 to obtain a score, with a range of 0 (extremely low functioning) to 100 (high functioning). Thus, a higher MDADI score represented better day-to-day functioning and better QOL.
Time Frame: Baseline and 5 years
Population: Of the 20 participants, 3 had progression of disease, and 2 were excluded due to insufficient survey compliance.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Reduced Dose Radiation | Standard Dose Radiation
Number analyzed (Participants) | 9 | 6
score on a scale | -8.12 (26.21) | -8.93 (18.31)

8. Secondary Outcome: Change in MD Anderson Symptom Inventory Symptom Inventory and Severity (MDASI-HN SI and SS)
Description: MD Anderson Symptom Inventory Symptom Inventory and Severity (MDASI-HN SI and SS) MDASI Head and Neck is a site-specific MDASI module which includes the core MDASI 13 symptom severity items (SS) and 6 symptom interference items (SI), alongside 9 items relevant to head and neck cancer. The scores are summed and a mean score is calculated on a scale of 0 (low severity or interference) to 10 (high severity or complete interference). In order to calculate the mean score, a majority of the subscale's items must have been completed.
  A lower or negative score reflects a better quality of life compared to baseline.
Time Frame: Baseline and 5 years
Population: Of the 20 participants, 3 had progression of disease, and 2 were excluded due to insufficient survey compliance.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Reduced Dose Radiation | Standard Dose Radiation
Number analyzed (Participants) | 9 | 6
score on a scale
  MDASI-HN SI | 0.64 (4.40) | 1.56 (1.92)
  MDASI-HN SS | 0.52 (2.11) | 1.48 (1.16)

9. Secondary Outcome: Change in Xerostomia Questionnaire (XQ)
Description: XQ is a nine questions survey developed specifically for xerostomia symptoms. The scores are summed and a mean score is calculated on a scale of 0 (low xerostomia interference) to 10 (high xerostomia interference). A lower or negative score reflects a better quality of life compared to baseline.
Time Frame: Baseline and 5 years
Population: Of the 20 participants, 3 had progression of disease, and 2 were excluded due to insufficient survey compliance.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Reduced Dose Radiation | Standard Dose Radiation
Number analyzed (Participants) | 9 | 6
score on a scale | 2.18 (4.07) | 4.38 (2.39)

10. Secondary Outcome: Change in European Organization for Research and Treatment of Cancer Questionnaire for Head and Neck (EORTC HN)
Description: The EORTC Head and Neck module was specifically designed and validated for head and neck cancer patients. This 35-item questionnaire contains 7 symptom scales (pain, swallowing, senses, speech, social eating, social contact, and sexuality), 6 single-item scales (difficulties of teeth, mouth opening, dry mouth, sticky saliva, coughing, and feeling ill), and 5 items about the additional use of pain medicine, nutritional supplements, and feeding tube and changes in body weight. All items were transformed to scales from 0 to 100, and divided into respective sub-scores of global health (GHS), functional (FS), and symptom scale (SS). Subscales from 0-100. A high score on global health and functional scale represents a better level of functioning, whereas a high score on a symptom scale and head and neck module indicates more severe symptoms.
Time Frame: Baseline and 5 years
Population: Of the 20 participants, 3 had progression of disease, and 2 were excluded due to insufficient survey compliance.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Reduced Dose Radiation | Standard Dose Radiation
Number analyzed (Participants) | 9 | 6
score on a scale
  EORTC GHS | 5.95 (27.52) | -30.56 (31.55)
  EORTC FS | 5.14 (30.38) | -6.33 (19.01)
  EORTC SS | -3.91 (22.36) | 14.97 (20.67)
  EORTC HN | -2.80 (20.55) | 8.97 (5.55)

ADVERSE EVENTS:
Time Frame: 5 years
Description: Adverse Events were not collected for the pre-randomization phase. Adverse events assessed for participants who were randomized.
Arm/Group | Pre-Randomization | Reduced Dose Radiation | Standard Dose Radiation
All-Cause Mortality (participants affected / at risk) | 0/0 | 2/12 | 1/8
Serious Adverse Events (participants affected / at risk) | 0/0 | 2/12 | 2/8
Other Adverse Events (participants affected / at risk) | 0/0 | 9/12 | 8/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pre-Randomization (N=0) | Reduced Dose Radiation (N=12) | Standard Dose Radiation (N=8)
Trigone oropharyngeal squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | NA | 0 | 1
Osteoradionecrosis (Musculoskeletal and connective tissue disorders) | NA | 0 | 1
Dental failure (Gastrointestinal disorders) | NA | 1 | 0
Oropharyngeal scarring and fibrosis (Injury, poisoning and procedural complications) | NA | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pre-Randomization (N=0) | Reduced Dose Radiation (N=12) | Standard Dose Radiation (N=8)
Mucositis (Gastrointestinal disorders) | NA | 1 | 1
Neutropenic fever (Infections and infestations) | NA | 0 | 1
Urinary retention (Renal and urinary disorders) | NA | 1 | 0
Acute hearing loss (Ear and labyrinth disorders) | NA | 1 | 0
Dehydration (Metabolism and nutrition disorders) | NA | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | NA | 1 | 1
Syncope (Cardiac disorders) | NA | 0 | 1
Opiod overdose (Injury, poisoning and procedural complications) | NA | 1 | 0
Hypothyroidism (Endocrine disorders) | NA | 6 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-02-21): https://cdn.clinicaltrials.gov/large-docs/39/NCT01706939/Prot_SAP_000.pdf